CLINICAL TRIAL: NCT05783362
Title: Pain Modulation Effectiveness: An Experimental Study Using Repeated Conditioned Pain Modulation as an Intervention and Analyzing Potential Predictors in Healthy Adults.
Brief Title: Pain Modulation Effectiveness (PME)
Acronym: PME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB202300187
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Healthy People

STUDY DESIGN:
Intervention Model Description: Individuals will be randomized to one of three groups: High Exposure (HE), Low Exposure (LE), No Exposure (NE).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Exposure (HE) (Experimental): Participants will receive five sessions total: four sessions of the Intervention, questionnaires, quantitative sensory testing, and CPM as an outcome in the first and fifth sessions.
  Interventions: Behavioral: Conditioned Pain Modulation (CPM)
- Low Exposure (LE) (Experimental): Participants will receive only two sessions in total: questionnaires, quantitative sensory testing, and CPM as an outcome at both sessions.
  Interventions: Behavioral: Conditioned Pain Modulation (CPM)
- No Exposure (NE) (No Intervention): This group controls for natural history response, and participants will receive two sessions of questionnaires, and CPM as an outcome, and quantitative sensory testing for one session (last session).

INTERVENTIONS:
Behavioral: Conditioned Pain Modulation (CPM) — Participants will receive a testing stimulus of pressure applied per ascending intensity at the web space of the foot until the pain reaches 40 out of 100, then discontinued. After testing the stimulus, participants will then receive a conditioning stimulus by immersing the non-dominant hand into the water-cooled by refrigeration unit with a temperature of 6 degree Celsius (males) or 8 degree Celsius (females) for 60 seconds. Subjects will be asked to rate the cold pain during the four 60-second trials. Participants completely removed their hand from the cold pressor for 30 seconds following each of the four 60-second immersions, during which time the testing stimulus will be re-applied per the sequential paradigm to the web space of the foot. Participants complete four 60-second periods of immersion. Conditioned pain modulation will be calculated as the average pain ratings of the second testing stimulus series minus the average pain ratings of the first testing stimulus series.
  Arms: High Exposure (HE); Low Exposure (LE)

SUMMARY:
Conditioned pain modulation (CPM) is the behavioral measure of diffuse noxious inhibitory control (DNIC), an endogenous pain inhibitory pathway in which pain inhibits pain. Conditioned pain modulation is less efficient in individuals with chronic pain conditions, and it is a predictor for the development of chronic pain. Continuous stimulation of central/cortical mechanisms through engaging CPM might alter pain processing and improve pain inhibition. Healthy participants will be randomly assigned to one of three groups: High Exposure (HE), Low Exposure (LE), and No Exposure (NE). Pre-and post-intervention pain sensitivity including conditioned pain modulation will be assessed. The study will assess the central pain modulatory mechanisms (measured by CPM) that have differential changes in participants who receive high exposure CPM as an intervention from those who receive low or no exposure. The study will also assess the magnitude and efficiency of CPM contributing additional variance to a regression model predicting pain sensitivity after positive and negative affect, pain anxiety, and depression are considered in the model, establishing measures of central pain processing, like CPM, as unique contributors to pain intensity.

DETAILED DESCRIPTION:
Background:

Pain is a widespread health condition that has a large burden on individuals, families, and society. Of the 39.4 million adults with pain that occurs most days and persists for more than three months, nearly two-thirds deem it "constantly present," and over half define it as "unbearable and excruciating". Pain may be classified as physiological and pathological. Nociceptive and inflammatory pain are physiological states that are protective and adaptive, whereas pathological pain is nonprotective and maladaptive.

The conditioned pain modulation (CPM) paradigm is a dynamic QST measure of a pain inhibitory process that lessens pain sensitivity in response to a remotely applied painful stimulus and is used to assess the ability of the person to endogenously inhibit pain. CPM may be a valuable tool in directing mechanistic-based approaches for treating painful conditions. For example, individuals with painful diabetic neuropathy and poorly functioning CPM have more significant analgesia when given duloxetine, a medication that augments conditioned pain modulation. Additionally, identifying and treating the source of pain is associated with positive changes in CPM. Healthy individuals demonstrate more efficient CPM when compared with people in pain and a systematic review of adults with chronic pain revealed that CPM efficiency improves after a reduction in pain. For example, total hip arthroplasty for treating painful osteoarthritis reduces pain and improves post-operative CPM. Collectively, these studies suggest that the CPM test has the potential to predict risk and treatment outcomes for chronic pain., therefore CPM may be considered an essential treatment moderator and mediator.

Activation of these central mechanisms (endogenous inhibitory systems) has also been proposed as the mechanism underpinning interventions used to treat various pain conditions. For example, evidence suggests that descending pain inhibitory systems (central mechanisms) play a fundamental role in mediating the analgesic effect of manipulation-induced pain modulation. Manual therapy activates afferent neuronal inputs that stimulate the central nervous system to inhibit pain through descending modulation. Like manual therapy, CPM inhibits pain through descending modulation. Continuous stimulation of central mechanisms through CPM should therefore alter pain processing and improve pain inhibition.

However, few studies have used CPM as an intervention, and none answer these research questions: 1) Does repeated exposure to conditioned pain modulation affect pain sensitivity? 2) Is analgesic efficacy of the nervous system predicted by the CPM effect? 3) Does CPM have therapeutic implications?

Understanding pain inhibitory mechanisms through this investigation would add further evidence to understanding the mechanism for chronic pain and might be a potential target for treating chronic pain.

Specific Aims:

Aim 1: To determine the extent to which repeated exposure to CPM protocols modifies pain sensitivity.

Hypothesis 1: CPM efficiency will increase in the high-exposure group compared to the low-exposure or No exposure group.

Aim 2: To determine the extent to which expectations affect the change in CPM efficiency.

Hypothesis 2: Participants with positive pain-related expectations will display a greater magnitude of improvement in CPM efficiency.

Research Plan:

The study in this proposal will be based on psychophysical data and self-reported questionnaires using methods approved by the University of Florida Institutional Review Board. This prospective experimental study involves participants without chronic pain conditions who will undergo baseline assessments, including psychological questionnaires and psychophysical approaches to measuring individual sensitivity and endogenous pain modulation. After an intervention period, participants will be reassessed. All assessments will be performed by an evaluator who will be blind to psychological measure data and group assignment.

Participants:

Seventy participants will be recruited by posted fliers approved by the IRB on the University of Florida campus and the Gainesville Florida community.

Inclusion criteria: a) Not currently seeking treatment for pain past month; b) between 18 - 75 years old.

Exclusion criteria: Participants will not be excluded based on race or gender but will be excluded if they meet any of the following a) non-English speaking; b) systemic medical condition is known to affect sensation (i.e., diabetes); c) regular use of prescription pain medication to manage pain; d) current or history of chronic pain condition; e) currently using blood thinning medication; f) any blood clotting disorder such as hemophilia; g) any contraindication to the application of ice or cold packs, such as uncontrolled hypertension, cold urticaria, cryoglobulinemia, paroxysmal cold hemoglobinuria, and circulatory compromise; h) involved in vigorous physical activities like heavy lifting, digging, aerobics or fast bicycling.

Recruitment and Informed Consent Procedure:

Potential participants interested in the study will respond to posted fliers and contact either the primary Investigator or co-investigator by phone or e-mail. The primary Investigator or co-investigator will read from an IRB-approved phone script or respond through an IRB-approved e-mail script to provide an overview of basic information about the study and answer questions. Participants wishing to participate will be scheduled for the formal consent process with either the Principal Investigator or co-investigator. Informed consent will occur in the Department of Physical Therapy lab space in the Health Science Center's Dental Wing. At that time, the primary Investigator or co-investigator will explain the study procedure, study purpose, benefits/risks of participating, and use of protected health information. The investigators will ensure appropriate time is spent with the participant to answer any questions and ensure he or she understands the procedures and risks associated with the study. If the participant chooses to participate, informed consent will be obtained from the participant as appropriate.

Measures:

Measures will be collected by the primary investigator, co-investigator, and/or research assistant under the direct supervision of the primary or co-investigator.

Questionnaires:

Demographic and Historical Factors:

Study participants will complete a standard intake information form including gender, age, employment status, marital status, educational level, and health history.

Expectation: Individuals will be asked what they expect exposure to the coldpressor task to do the amount of pressure needed to generate pain (see "Intervention" for the coldpressor task).

Quantitative Sensory Testing:

Conditioned Pain Modulation (as an assessment): Participants will receive a testing stimulus of pressure applied to the web space of the dominant foot. Pressure will be applied per ascending intensity until the pain reaches 40 out of 100, then discontinued. Participants are instructed to say "stop" or "pain" so the stimulus can be terminated "when you feel pain equal to 40 out of 100." Participants will then receive a conditioning stimulus contact heat stimulus applied to the thenar of the left hand for 60 s at an intensity of 46.5 ◦C (Matre, 2013). Subjects will be asked to rate the heat pain and unpleasantness during a 60-second trial. Subjects will be instructed that they may remove their hand at any time if the heat is intolerable. After 60 seconds, the contact heat will be completely removed, and the testing stimulus will be re-applied to the web space of the dominant foot. Conditioned pain modulation will be calculated as the average pain ratings of the second testing stimulus series minus the average pain ratings of the first testing stimulus series. Negative numbers indicate efficient pain modulation.

Procedure:

Participants who consent will sign up for individual blocks of testing time (90 minutes) to take part in the experiment. Participants who consent will sign up for individual blocks of testing time (90 minutes) to take part in the experiment. Participants will complete expectation questions before every protocol session. Blood pressure will be assessed with a digital blood pressure monitor before every session. If blood pressure exceeds 140/90 mmHg, the participant will be removed from the study session and notified of the blood pressure reading. Next, a baseline assessment of pain sensitivity will be completed. After testing, participants sit quietly for 15 minutes to allow changes in pain sensitivity to normalize after pre-intervention CPM testing (Lewis et al., 2012). Individuals will be randomized to one of three groups: High Exposure (HE), Low Exposure (LE), No Exposure (NE).

High Exposure: Participants will receive five sessions total: four sessions of the Intervention, questionnaires, quantitative sensory testing, and CPM as an outcome in the first and fifth sessions.

Low Exposure: Participants will receive only two sessions in total: questionnaires, quantitative sensory testing, and CPM as an outcome at both sessions.

No Exposure: This group controls for natural history response, and participants will receive two sessions of questionnaires, and CPM as an outcome, and quantitative sensory testing for one session (last session).

High exposure group will be attending 5 sessions (about once every 72 hours) for two weeks. The other two groups (Low Exposure and No Exposure) come twice (the second visit about 2 weeks later). Visits can last 1 to 1.5 hours.

Intervention:

CPM: Participants will receive a testing stimulus of pressure applied to the web space of the dominant foot. Pressure is applied per ascending intensity until the pain reaches 40 out of 100, then discontinued. Participants will be instructed to say "stop" or "pain" so the stimulus can be terminated "when you feel pain equal to 40 out of 100." This will be repeated twice, and the average will be analyzed (Yarnitsky et al., 2015). Participants will then receive a conditioning stimulus by immersing non-dominant hand into the water cooled by a refrigeration unit (NESLAB RTE 7 Digital One, Thermo Scientific Co., Massachusetts, USA) that circulates water continuously to maintain a constant temperature of six degree Celsius (males) or eight degree Celsius (females) for 60 seconds. Subjects will be asked to rate the cold pain and unpleasantness during the four 60-second trials. Subjects will be instructed that they may remove their hand at any time if the water is intolerable. If this occurs, or if subjects rate the pain higher than 50 (0-100 scale), the bath temperature will be increased for the subsequent trial. If the ratings are less than 20, a small about of ice was added to lower the temperature by up to 4o Celsius. Participants completely removed their hand from the cold pressor for 30 seconds following each of the four 60-second immersions, during which time the testing stimulus will be re-applied per the sequential paradigm to the web space of the foot. Participants complete four 60-second periods of immersion. Conditioned pain modulation will be calculated as the average pain ratings of the second testing stimulus series minus the average pain ratings of the first testing stimulus series. Negative numbers indicate efficient pain modulation.

Immediately following the assigned intervention, pain sensitivity measures will be re-assessed as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Not currently seeking treatment for pain past month;
2. between 18 - 75 years old.

Exclusion Criteria: Participants will not be excluded based on race or gender but will be excluded if they meet any of the following

1. non-English speaking;
2. systemic medical condition is known to affect sensation (i.e., diabetes);
3. regular use of prescription pain medication to manage pain;
4. current or history of chronic pain condition;
5. currently using blood thinning medication;
6. any blood clotting disorder such as hemophilia;
7. any contraindication to the application of ice or cold packs, such as uncontrolled hypertension, cold urticaria, cryoglobulinemia, paroxysmal cold hemoglobinuria, and circulatory compromise;
8. involved in vigorous physical activities like heavy lifting, digging, aerobics or fast bicycling.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Conditioned Pain Modulation as an assessment | Two weeks
  Participants will receive a testing stimulus of pressure applied per ascending intensity at the web space of the foot until the pain reaches 40 out of 100, then discontinued. After testing the stimulus, Participants will receive a conditioning stimulus contact heat stimulus applied to the thenar of the left hand for 60 s at an intensity of 46.5 ◦C. Subjects will be asked to rate the heat pain during the four 60-second trials. Subjects will be instructed that they may remove their hand at any time if the heat is intolerable. After 60 seconds, the contact heat will be completely removed, and the testing stimulus will be re-applied to the web space of the dominant foot. Conditioned pain modulation will be calculated as the average pain ratings of the second testing stimulus series minus the average pain ratings of the first testing stimulus series. Negative numbers indicate efficient pain modulation
Expectations | Two Weeks
  Individuals will be asked what they expect exposure to the coldpressor task to do the amount of pressure needed to generate pain (see "Intervention" for the coldpressor task).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bishop, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cruz-Almeida Y, Fillingim RB. Can quantitative sensory testing move us closer to mechanism-based pain management? Pain Med. 2014 Jan;15(1):61-72. doi: 10.1111/pme.12230. Epub 2013 Sep 6. PMID 24010588
- [Background] Damien J, Colloca L, Bellei-Rodriguez CE, Marchand S. Pain Modulation: From Conditioned Pain Modulation to Placebo and Nocebo Effects in Experimental and Clinical Pain. Int Rev Neurobiol. 2018;139:255-296. doi: 10.1016/bs.irn.2018.07.024. Epub 2018 Aug 14. PMID 30146050
- [Background] Fong A, Schug SA. Pathophysiology of pain: a practical primer. Plast Reconstr Surg. 2014 Oct;134(4 Suppl 2):8S-14S. doi: 10.1097/PRS.0000000000000682. PMID 25255013
- [Background] Goldberg DS, McGee SJ. Pain as a global public health priority. BMC Public Health. 2011 Oct 6;11:770. doi: 10.1186/1471-2458-11-770. PMID 21978149
- [Background] Goubert D, Danneels L, Cagnie B, Van Oosterwijck J, Kolba K, Noyez H, Meeus M. Effect of Pain Induction or Pain Reduction on Conditioned Pain Modulation in Adults: A Systematic Review. Pain Pract. 2015 Nov;15(8):765-77. doi: 10.1111/papr.12241. Epub 2014 Nov 11. PMID 25387406
- [Background] Ibancos-Losada MDR, Osuna-Perez MC, Castellote-Caballero MY, Diaz-Fernandez A. Conditioned Pain Modulation Effectiveness: An Experimental Study Comparing Test Paradigms and Analyzing Potential Predictors in a Healthy Population. Brain Sci. 2020 Aug 30;10(9):599. doi: 10.3390/brainsci10090599. PMID 32872642
- [Background] Kennedy J, Roll JM, Schraudner T, Murphy S, McPherson S. Prevalence of persistent pain in the U.S. adult population: new data from the 2010 national health interview survey. J Pain. 2014 Oct;15(10):979-84. doi: 10.1016/j.jpain.2014.05.009. PMID 25267013
- [Background] Kosek E, Ordeberg G. Abnormalities of somatosensory perception in patients with painful osteoarthritis normalize following successful treatment. Eur J Pain. 2000;4(3):229-38. doi: 10.1053/eujp.2000.0175. PMID 10985866
- [Background] Nir RR, Granovsky Y, Yarnitsky D, Sprecher E, Granot M. A psychophysical study of endogenous analgesia: the role of the conditioning pain in the induction and magnitude of conditioned pain modulation. Eur J Pain. 2011 May;15(5):491-7. doi: 10.1016/j.ejpain.2010.10.001. Epub 2010 Oct 28. PMID 21035364
- [Background] Nir RR, Yarnitsky D. Conditioned pain modulation. Curr Opin Support Palliat Care. 2015 Jun;9(2):131-7. doi: 10.1097/SPC.0000000000000126. PMID 25699686
- [Background] Pud D, Granovsky Y, Yarnitsky D. The methodology of experimentally induced diffuse noxious inhibitory control (DNIC)-like effect in humans. Pain. 2009 Jul;144(1-2):16-9. doi: 10.1016/j.pain.2009.02.015. Epub 2009 Apr 8. No abstract available. PMID 19359095
- [Background] Yarnitsky D. Conditioned pain modulation (the diffuse noxious inhibitory control-like effect): its relevance for acute and chronic pain states. Curr Opin Anaesthesiol. 2010 Oct;23(5):611-5. doi: 10.1097/ACO.0b013e32833c348b. PMID 20543676
- [Background] Yarnitsky D, Bouhassira D, Drewes AM, Fillingim RB, Granot M, Hansson P, Landau R, Marchand S, Matre D, Nilsen KB, Stubhaug A, Treede RD, Wilder-Smith OH. Recommendations on practice of conditioned pain modulation (CPM) testing. Eur J Pain. 2015 Jul;19(6):805-6. doi: 10.1002/ejp.605. Epub 2014 Oct 20. PMID 25330039
- [Background] Yarnitsky D, Granot M, Nahman-Averbuch H, Khamaisi M, Granovsky Y. Conditioned pain modulation predicts duloxetine efficacy in painful diabetic neuropathy. Pain. 2012 Jun;153(6):1193-1198. doi: 10.1016/j.pain.2012.02.021. Epub 2012 Apr 3. PMID 22480803
- [Background] 15. Souvlis, T., Vicenzino, B., and Wright. A. (2004). Neurophysiological effect of spinal manual therapy. Grieve's Modern Manual Therapy: The Vertebral Column. Edited by Jeffrey D. Boyling and Gwendolen A. Jull. Edinburgh, United Kingdom: Churchill Livingstone.367-380.
- [Derived] Rana P, Robinson ME, Alappattu MJ, Riley Iii J, Lott D, Bishop MD. Impact of repeated exposure to CPM on CPM efficiency and pain sensitivity in healthy adults: a randomized controlled trial. Front Pain Res (Lausanne). 2025 Nov 13;6:1677563. doi: 10.3389/fpain.2025.1677563. eCollection 2025. PMID 41322117